CLINICAL TRIAL: NCT06733350
Title: Investigating the Effect of Testosterone Replacement Therapy Among Hypogonadal Men With Localized Prostate Cancer on Active Surveillance
Brief Title: Testosterone Replacement Therapy for the Treatment of Low Testosterone in Hypogonadal Men With Localized Prostate Cancer on Active Surveillance
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Implementation issues
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I-3920923; NCI-2024-09551 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I-3920923 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Localized Prostate Carcinoma; Stage I Prostate Cancer AJCC v8; Stage II Prostate Cancer AJCC v8; Stage III Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Specimen Handling; Magnetic Resonance Spectroscopy; Watchful Waiting; Observation; Testosterone Propionate; Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group 1 (AS) (Active Comparator): Patients with normal testosterone level undergo standard AS for up to 5 years in the absence of disease progression. Patients undergo blood sample collection and MRI throughout the trial and may undergo prostate biopsy on study.
  Interventions: Procedure: Biopsy of Prostate; Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Imaging; Other: Patient Observation; Other: Questionnaire Administration
- Group 2 (TRT, AS) (Experimental): Patients with low testosterone level associated with hypogonadal symptoms and willing to receive TRT receive testosterone per treating physician discretion via injection, gel, lotion, or transdermal patch and undergo standard AS for up to 5 years in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection and MRI throughout the trial and may undergo prostate biopsy on study.
  Interventions: Procedure: Biopsy of Prostate; Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Imaging; Other: Patient Observation; Other: Questionnaire Administration; Drug: Therapeutic Testosterone
- Group 3 (AS) (Active Comparator): Patients with low testosterone level with no symptoms, or low testosterone level associated with hypogonadal symptoms but declined TRT undergo standard AS for up to 5 years in the absence of disease progression. Patients undergo blood sample collection and MRI throughout the trial and may undergo prostate biopsy on study.
  Interventions: Procedure: Biopsy of Prostate; Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Imaging; Other: Patient Observation; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biopsy of Prostate — Undergo prostate biopsy
  Other Names: Prostate Biopsy; Prostatic Biopsy
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Patient Observation — Undergo standard AS
  Other Names: Active Surveillance; deferred therapy; expectant management; Observation; Watchful Waiting
Other: Questionnaire Administration — Ancillary studies
Drug: Therapeutic Testosterone — Given via injection, gel, lotion, or transdermal patch
  Other Names: Mertestate; Testoderm; Testolin; Testosterone; Testostroval; Testostroval-PA; Testro AQ; Trans-Testosterone; Virosterone
  Arms: Group 2 (TRT, AS)

SUMMARY:
This phase IV trial studies the effects of testosterone replacement therapy (TRT) on treatment outcomes in hypogonadal men with prostate cancer that has not spread to other parts of the body (localized) and who are on active surveillance (AS). AS in prostate cancer involves closely watching the patient's condition through regular physical exams and blood tests, but not giving treatment unless there are changes in test results. It can be a practical alternative to treatment in localized prostate cancer. Hypogonadal men have low testosterone associated with symptoms such as low libido and erectile problems. TRT can be used to treat hypogonadism by increasing testosterone levels, which may improve associated symptoms. TRT is often not used in men with prostate cancer due to concerns it may lead to the cancer growing or spreading. This may lead hypogonadal men to have a poor quality of life or to discontinue AS. TRT may improve treatment and quality of life outcomes in hypogonadal men with localized prostate cancer on active surveillance.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To investigate the impact of TRT on Gleason grade progression in hypogonadal men with localized prostate cancer on active surveillance, and the association between TRT and the likelihood of discontinuation of active surveillance in the same population.

II. To assess the impact of TRT on the quality of life, including changes in the International Prostate Symptom Score (IPSS) and the association with sexual health measured by the Sexual Health Inventory for Men (SHIM), in hypogonadal men with localized prostate cancer on active surveillance.

SECONDARY OBJECTIVES:

I. To examine the influence of TRT on radiographic progression in hypogonadal men with localized prostate cancer on active surveillance, by assessing changes in the size of abnormal magnetic resonance imaging (MRI) lesions.

II. To evaluate the association between TRT and biochemical progression by analyzing changes in prostate-specific antigen (PSA) levels over time in the studied population.

III. To systematically monitor and document TRT-related adverse events and complications, and concurrently assess the association between TRT and the likelihood of discontinuation due to adverse events in the studied population.

OUTLINE: Patients are assigned to 1 of 3 groups.

GROUP 1: Patients with normal testosterone level undergo standard AS for up to 5 years in the absence of disease progression. Patients undergo blood sample collection and MRI throughout the trial and may undergo prostate biopsy on study.

GROUP 2: Patients with low testosterone level associated with hypogonadal symptoms and willing to receive TRT receive testosterone per treating physician discretion via injection, gel, lotion, or transdermal patch and undergo standard AS for up to 5 years in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection and MRI throughout the trial and may undergo prostate biopsy on study.

GROUP 3: Patients with low testosterone level with no symptoms, or low testosterone level associated with hypogonadal symptoms but declined TRT undergo standard AS for up to 5 years in the absence of disease progression. Patients undergo blood sample collection and MRI throughout the trial and may undergo prostate biopsy on study.

ELIGIBILITY:
Inclusion Criteria:

* Men aged ≥ 18 years
* Men with localized prostate cancer are eligible for active surveillance (National Comprehensive Cancer Network [NCCN] very low, low, and intermediate favorable risk group)
* Participant must understand the investigational nature of this study and sign an independent ethics committee/institutional review board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Patients with NCCN intermediate unfavorable, high risk, or very high-risk localized prostate cancer
* Patients with contraindications to TRT, which include,

  * Locally advanced or metastatic prostate cancer
  * Male breast cancer
  * Men with an active desire to have children
  * Hematocrit levels > 54% or baseline hematocrit of 48-50%
  * Uncontrolled or poorly controlled congestive heart failure
  * IPSS score > 19
  * Family history of venous thromboembolism
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to participate in the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2029-01-15 (Estimated); Study Completion 2029-01-15 (Estimated)

PRIMARY OUTCOMES:
Gleason grade progression | From start of active surveillance until any progression in primary, secondary, or a combination of Gleason grades, definitive treatment, or last follow-up, assessed up to 5 years
  The Gleason grade progression will be summarized by group using standard Kaplan-Meier methods, where estimates of the median or specified rates will be obtained. Comparisons will be made between groups using the log-rank test. As exploratory analyses, Cox regression models may be considered to adjust for relevant demographic or clinical confounders. The Bonferroni method will be used to control the family-wise error rate at 0.10.
Discontinuation of active surveillance | From start of active surveillance until discontinuation of active surveillance due to any cause or last follow-up, assessed up to 5 years
  The discontinuation of active surveillance will be summarized by group using standard Kaplan-Meier methods, where estimates of the median or specified rates will be obtained. Comparisons will be made between groups using the log-rank test. As exploratory analyses, Cox regression models may be considered to adjust for relevant demographic or clinical confounders. The Bonferroni method will be used to control the family-wise error rate at 0.10.
International Prostate Symptom Score (Quality-of-life) | Up to 5 years
  Will be modeled as a function of group, timepoint, their two-way interaction, and a random subject effect using linear mixed models. Tests about the appropriate contrasts of model estimates will be used to compare mean changes in quality of life between groups at specified timepoints. All model assumptions will be verified graphically, and transformations applied as appropriate. As exploratory analyses, additional models may be considered to adjust for relevant demographic or clinical confounders. The Bonferroni method will be used to control the family-wise error rate at 0.10.
Sexual Health Inventory for Men score (Quality-of-life) | Up to 5 years
  Will be modeled as a function of group, timepoint, their two-way interaction, and a random subject effect using linear mixed models. Tests about the appropriate contrasts of model estimates will be used to compare mean changes in quality of life between groups at specified timepoints. All model assumptions will be verified graphically, and transformations applied as appropriate. As exploratory analyses, additional models may be considered to adjust for relevant demographic or clinical confounders. The Bonferroni method will be used to control the family-wise error rate at 0.10.

SECONDARY OUTCOMES:
Radiographic progression | From start of active surveillance until radiographic progression, definitive treatment, or last follow-up, assessed up to 5 years
  Will assess change in the size of abnormal magnetic resonance imaging (MRI) lesions, if any. Will utilize the PRECISE scoring system, which considers factors such as changes in lesion volume or appearance on MRI and can provide a standardized and objective method for assessing progression. Will be summarized by group using standard Kaplan-Meier methods, where estimates of the median or specified rates will be obtained. Comparisons will be made between groups using the log-rank test.
Biochemical progression | From the start of active surveillance until prostate specific antigen (PSA) progression, definitive treatment, or last follow-up, assessed up to 5 years
  Will be assessed by change in the PSA over time. Will be summarized by group using standard Kaplan-Meier methods, where estimates of the median or specified rates will be obtained. Comparisons will be made between groups using the log-rank test.
Incidence of testosterone replacement therapy (TRT)-related adverse events | Up to 5 years
  Will be assessed in Group 2 patients. Will be summarized by attribution and grade using frequencies and relative frequencies.
Incidence of TRT-related complications | Up to 5 years
  Will be assessed in Group 2 patients. Will be summarized by attribution and grade using frequencies and relative frequencies.
TRT discontinuation | Up to 5 years
  Will be assessed in Group 2 patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Aly, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States